CLINICAL TRIAL: NCT06738667
Title: Study on Imaging Characteristics and Predictive Radiology of Brain Network Regulation by Acupuncture in Patients with Painful Temporomandibular Disorders
Brief Title: Acupuncture for Painful Temporomandibular Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Li bin, Professor, Beijing Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SL-2024BL02-100-02
Record Dates: First submitted 2024-12-06; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Temporomandibular Disorders (TMD)
Keywords: Temporomandibular disorders; Acupuncture; Magnetic resonance imaging; Randomized controlled trial; Protocol
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- acupuncture (Experimental): Patients in the acupuncture group will receive treatment at specified acupoints, performed by acupuncturists with at least five years of experience. The acupoints include bilateral Hegu (LI4), Yanglingquan (GB34), and affected-side Jiache (ST6), Xiaguan (ST7), and Tinggong (SI19).
  Interventions: Other: Acupuncture
- sham acupuncture (Sham Comparator): Patients in the sham group will receive noninvasive acupuncture at the same acupoints as the acupuncture group. Sham needles, which resemble real needles but are blunt and slide within their handles, will be applied using the Park Sham device, secured to the skin with a self-adhesive pad. The procedure of manipulation is the same as for acupuncture, but without Deqi.
  Interventions: Other: Sham treatment

INTERVENTIONS:
Other: Acupuncture — Patients in the acupuncture group will receive treatment at specified acupoints, performed by acupuncturists with at least five years of experience. The acupoints include bilateral Hegu (LI4), Yanglingquan (GB34), and affected-side Jiache (ST6), Xiaguan (ST7), and Tinggong (SI19). Participants will lie supine, and the skin will be sterilized. Sterile stainless-steel needles (0.25 mm diameter, 40 mm length) will be inserted using a guide device and a self-adhesive pad. Needles will be manipulated for at least 10 seconds to induce Deqi. Participants will receive 30 minutes of acupuncture for twelve sessions (3 per week for 4 weeks).
  Arms: acupuncture
Other: Sham treatment — The Park Sham device will be used for the sham acupuncture group. To maintain blinding, the acupuncture ritual will be identical in both groups, with the following exceptions: patients in the sham group will receive noninvasive acupuncture at the same acupoints as the acupuncture group. Sham needles, which resemble real needles but are blunt and slide within their handles, will be applied using the Park Sham device, secured to the skin with a self-adhesive pad. The procedure of manipulation is the same as for acupuncture, but without Deqi.
  Arms: sham acupuncture

SUMMARY:
Temporomandibular disorder (TMD) is a common musculoskeletal pain condition affecting the jaw, and acupuncture is often used for treatment, though its neurological mechanisms are unclear. This study investigates the neural mechanisms of acupuncture in TMD using functional MRI (fMRI), structural MRI (sMRI), and diffusion tensor imaging (DTI), alongside machine learning to predict treatment outcomes. This study aims to enhance understanding of acupuncture's effects on TMD and improve personalized treatment approaches.

DETAILED DESCRIPTION:
A randomized, single-blind, sham-controlled trial will enroll 48 patients, divided into acupuncture and sham acupuncture groups. The study will consist of a 1-week baseline, 4-week treatment, and 8-week follow-up period, with 30-minute sessions three times a week for 12 sessions. Primary outcomes include changes in Visual Analog Scale (VAS) scores at week 4, with secondary outcomes including VAS changes at week 8, jaw function, and scores on pain, sleep, and mental health scales. Multimodal MRI scans will assess brain changes at baseline, post-treatment, and follow-up. Our research is a randomized controlled trial (RCT) combining sMRI, fMRI, and DTI to explore the efficacy of acupuncture in TMD treatment, using multi-modal imaging to provide a comprehensive biological profile of TMD patients. Our study aims to (1) analyze brain structural and functional network changes post-acupuncture, explore the relationship between central imaging and clinical symptom changes, and (2) predict individual treatment outcomes for TMD.

ELIGIBILITY:
Inclusion Criteria:

1. Having a history of pain-related TMD for at least three months;
2. Aged between 18 and 70 years;
3. Voluntary participation in the trial with signed informed consent.

Exclusion Criteria:

1. Having received occlusal splint, injection therapy, acupuncture, biofeedback, transcutaneous nerve stimulation, or TMD-specific medication (e.g., corticosteroids, benzodiazepines, sedative hypnotics, muscle relaxants, opioids, antidepressants, or anticonvulsants) for managing facial pain within one month before the screening period;
2. Having suffered from pain of dental origin, trauma, sinus pathology, neuropathic origin, inflammatory systemic diseases and cancer;
3. Having a history of rheumatoid arthritis;
4. Presence of mental illness or substance abuse;
5. Pregnant, lactating, or planning to become pregnant;
6. Participants with common contra-indications for MRI such as claustrophobia or metal implants.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | From baseline (week 0) to the end of treatment (week 4) and the end of follow-up period (week 16)
  The VAS is a self-administered instrument, ranging from 0 (no pain at all) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
Magnetic Resonance Imaging | From baseline (week 0) to the end of treatment (week 4) and the end of follow-up period (week 16)
  (1) structural MRI (sMRI): voxel-based whole-brain voxel-mirrored homotopic connectivity (VMHC), cortical thickness, gray matter volume (GMV), white matter volume (WMV), total brain volume (TBV); (2) fMRI: independent component analysis (ICA)-based functional connectivity (FC), seed-based FC, amplitude of low-frequency fluctuation (ALFF), fractional ALFF, regional homogeneity (ReHo), degree centrality (DC); (3) DTI: mean diffusivity (MD), radial diffusivity (RD), axial diffusivity (AD), and fractional anisotropy (FA).
Effective response rate | From baseline (week 0) to the end of treatment (week 4) and the end of follow-up period (week 16)
  Effective response rate is revealed as proportion of participants whose average VAS scores decrease by at least 30% or 50%.
Jaw Opening and Movement | From baseline (week 0) to the end of treatment (week 4) and the end of follow-up period (week 16)
  It is an evaluation of physical function, including 6 items: pain-free jaw opening (mm), maximum unassisted jaw opening (mm), maximum assisted jaw opening (mm), left lateral movement (mm), right lateral movement (mm), and protrusion movement (mm).
Graded Chronic Pain Scale | From baseline (week 0) to the end of treatment (week 4) and the end of follow-up period (week 16)
  GCPS assesses disability, pain intensity, and whether an individual can work due to pain. It comprises three items for pain intensity, four items for function, and one item for the number of days with pain. Each item is scored on a scale of 0-10, higher scores indicate greater pain.
Jaw Function Limitation Scale-20 | From baseline (week 0) to the end of treatment (week 4) and the end of follow-up period (week 16)
  JFLS-20 is an organ-specific instrument that assesses the functional status of the masticatory system. It includes 20 items across 3 domains, with responses for each functional item ranging from 0 (no limitation) to 10 (severe limitation).
Depression Anxiety and Stress Scale-21 | From baseline (week 0) to the end of treatment (week 4) and the end of follow-up period (week 16)
  DASS-21 is used to measure emotional states. It consists of three independent subscales with a total of 21 items, with seven items each for depression, anxiety, and stress subscales. Each item is assessed using a Likert scale (0 = did not apply to me at all, 3 = applied to me very much, or most of the time). A higher score indicates greater severity of emotional distress
Pittsburgh Sleep Quality Index | From baseline (week 0) to the end of treatment (week 4) and the end of follow-up period (week 16)
  PSQI evaluates participants' sleep quality and disturbances over the preceding month. It consists of 19 items, including 4 open questions and 15 Likert-type questions, each scored on a scale from 0 to 3. These 19 items are organized into seven component scores. Higher scores reflect more severe sleep disturbances, with a cutoff score of 5 indicating poor sleep quality.
Pressure Pain Threshold | From baseline (week 0) to the end of treatment (week 4)
  PPT will be measured at five points: masseter, temporalis, sternocleidomastoid, trapezius, and TMJ, using a pressure algometer (Somedic AB, Sweden). Each measurement point will be assessed three times, with a two-minute interval between measurements. The lowest value from each point will be recorded by a trained assessor, and the final value will represent the average of the three measurements. Lower PPT values indicate greater pain sensitivity.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital of Traditional Chinese Medicine, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No